CLINICAL TRIAL: NCT02530086
Title: Prospective Study of Non-operative Management of SBO Without Nasogastric Tube Placement
Acronym: NoNGT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was closed due to lack of personnel for recruitment/enrollment purposes.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1504015652
Record Dates: First submitted 2015-08-17; First posted 2015-08-20 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Small Bowel Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placement of a Nasogastric tube (Active Comparator): Placement of a Nasogastric tube
  Interventions: Procedure: Nasogastric tube placement
- No placement of a Nasogastric tube (Experimental): No placement of a Nasogastric tube
  Interventions: Procedure: No Nasogastric tube use

INTERVENTIONS:
Procedure: Nasogastric tube placement — Placement of a Nasogastric tube
  Arms: Placement of a Nasogastric tube
Procedure: No Nasogastric tube use — No placement of a Nasogastric tube
  Arms: No placement of a Nasogastric tube

SUMMARY:
A prospective randomized trial comparing non-operative management of small bowel obstruction due to adhesions with or without a naso-gastric tube (NGT).

DETAILED DESCRIPTION:
The study will be conducted in a prospective randomized design using the patient population admitted to any of the general surgery services at Yale New Haven Hospital and presenting with the presumed diagnosis of adhesive small bowel obstruction (SBO) to Yale New Haven Hospital. All patients will be at least 30 days from any prior abdominal operative procedure. Diagnosis of SBO will be by CT scan of the abdomen thereby excluding patients with obstruction due to incarcerated hernias and minimizing the possibility the obstruction is due to malignancy, volvulus or other cause. All patients selected for non-operative management by the attending physician will be eligible for randomization to either the "Nasogastric Tube Decompression" or "No Decompression" groups. Eligible patients will be within 6 hours of hospital admission and not have had a naso-gastric tube (NGT) placed. Patients who have a NGT placed by emergency physicians prior to consultation to the emergency general surgery will be excluded. Patients who require NGT placement prior to being approached for enrollment or prior to randomization will, if agreeable, be enrolled in a prospective observational group of patients that will have the same data elements collected.

Study Procedures:

Randomization:

Once consent from the patient or his/her surrogate has been obtained, eligible patients will be randomized to either the "Nasogastric Tube Decompression" or the "No Decompression" group. Sequentially numbered opaque sealed envelopes will be maintained in the locked office of the surgical critical care fellow in the surgical intensive care unit. The grouping assignment within these envelopes will be generated from computerized random number tables. Patients randomized to nasogastric decompression will have a NGT placed within one hour of randomization.

Patient Management:

If patients in the "No Decompression" group develop recurrent or intractable emesis unresponsive to anti-emetic medication or are deemed unsafe to be trialed with anti-emetic medication due to a change in mental status by the attending physician they will have an NGT placed and they will be followed as a third group of patients that failed management without NGT decompression. Recurrent and/or intractable emesis will be defined as two or more episodes of emesis of at least 50cc within a twelve hour period or a single large volume emesis of 300cc or more.

For these patients NGT placement will not be mandatory however if patients do develop this volume of emesis NGT placement will be considered consistent with the protocol. Change in mental status will be loosely defined as the deterioration of the Glasgow Coma Scale (GCS) to less than 14, however this will remain at the discretion of the attending physician. For patients that have failure of NGT placement they will be managed at the discretion of the attending surgeon but analyzed using an intention to treat methodology.

All other standard care for patients with SBO including intravenous fluids, correction of electrolytes and management of chronic medical problems will be at the discretion of the attending surgeon. All patients will be monitored daily with clinical examination for the development of complications (vomiting, worsening abdominal pain, abnormal vital signs, leukocytosis, fevers). Patients' subjective comfort levels will also be assessed daily in each group using a visual analog scale. Pain will be managed will be with IV morphine unless an allergy is present or develops in which case an alternative narcotic will be used based on the decision of the treating physician. Improvement will be followed by return of bowel function, improving abdominal pain and resolution of symptoms. The time taken to resolution of symptoms in each group will be followed, as well as the relative number of patients improving and deteriorating. All care decisions beyond the initial NGT placement, choice of anti-emetic and choice of analgesic will be at the discretion of the attending surgeon. These decisions may include but are not limited to NGT placement and removal, laboratory testing, imaging (Abdominal X-rays and/or CT scan), diet advancement, and need for operative intervention.

Should a patient chose to withdraw from the study at any point after randomization management of the NGT will then also come within the purview of the attending physician. This may include placement of a NGT if the patient had been randomized to the no NGT arm or removal even if in the NGT was placed as part of the protocol.

Primary Outcomes:

1. Hospital length of stay

Secondary Outcomes

1. Pain level, as measured by the visual analog scale and documented by the treating nurse. The maximum and mean score for each day will be recorded. Pain will also be assessed by the amount of used.
2. Duration of NGT use in hours.
3. The number of abdominal and chest imaging tests prior to discharge or operation whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients over 18 years of age who meet the following criteria will be recruited if identified:

  * Admitted to a general surgery service with a presumptive diagnosis of adhesive SBO with or without a history of abdominal surgery. Have had no abdominal surgery in the 30 days prior to enrollment.
  * Present from home or a long term care facility.
  * CT scan of the abdomen performed within 36 hours of admission consistent with small bowel obstruction and without evidence the obstruction is due to an incarcerated hernia, malignancy or volvulus.
  * Planned attempt at non-operative management by the attending surgeon.
  * Have the capacity to provide informed consent for themselves.

Exclusion Criteria:

* Patient is deemed to need operative intervention at the time of presentation
* Pregnancy
* Contra-indication to NGT insertion
* Presence of a gastric feeding tube or dependent on tube feeding or parenteral nutrition on admission.
* Inability of the patient to protect their airway should emesis occur (as judged by the attending surgeon).
* Intractable emesis on admission.
* Abdominal surgery within 30 days prior to admission.
* Patients transferred from an inpatient status at another acute care hospital will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay | 30 days
  Total hospital length of stay.

SECONDARY OUTCOMES:
Pain measured on a visual analogue scale | 30 days
  Pain will be measured daily using a visual analog scale and milligrams of morphine used.
Duration of nasogastric decompression | 30 days
Number of radiographic studies ordered | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Schuster, MD, MPH, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States